CLINICAL TRIAL: NCT03421652
Title: Phase II Trial of Concurrent Nivolumab in Urothelial Bladder Cancer With Radiation Therapy in Localized/Locally Advanced Disease for Chemotherapy Ineligible Patients [NUTRA]
Brief Title: Nivolumab and RT in Treating Patients With Localized/Locally Advanced Urothelial Bladder Cancer Ineligible for Chemo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Nitin Vaishampayan, MD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-195
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Stage II Bladder Urothelial Carcinoma AJCC v6 and v7; Stage III Bladder Urothelial Carcinoma AJCC v6 and v7; Stage IV Bladder Urothelial Carcinoma AJCC v7
MeSH Terms: interventions — Nivolumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, radiation therapy) (Experimental): Given IV
  Interventions: Drug: Nivolumab; Radiation: Radiation

INTERVENTIONS:
Drug: Nivolumab — Patients receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 14 days (2 weeks) for up to 14 courses (6 months) in the absence of disease progression or unacceptable toxicity. Beginning 3 days of course 1, patients undergo radiation therapy over 32-35 on weeks 1, 3, 5, 7 and 9.
  Other Names: 946414-94-4; BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Radiation — Beginning 3 days of course 1, patients undergo radiation therapy over 32-35 on weeks 1, 3, 5, 7 and 9.

SUMMARY:
This phase II trial studies how well nivolumab works with radiation therapy in treating patients with urothelial bladder cancer that has spread from its original site of growth to nearby tissues or lymph nodes and are ineligible for chemotherapy. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving nivolumab and radiation therapy may work better in treating patients with urothelial bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the 12-month rate of progression-free survival (PFS) achieved with the combination of nivolumab, a programmed death (PD-1) inhibitor, and radiation therapy in localized/locally advanced urothelial cancer patients, who are chemotherapy ineligible, to a historical control reference 12-month PFS rate.

SECONDARY OBJECTIVES:

I. To assess the toxicity of concurrent nivolumab and radiation therapy in urothelial cancer.

II. To determine overall response rate (ORR). III. To determine metastasis-free survival (MFS). IV. To determine overall survival (OS). V. To evaluate the quality of life and bladder functioning during and after the therapy.

VI. To explore the relationships of PD-1 expression, PDL-1 expression, and the Th1/Th2 cytokine ratio to clinical outcomes (response, PFS, MFS, and OS).

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 14 days (2 weeks) for up to 14 courses (6 months) in the absence of disease progression or unacceptable toxicity. Beginning 3 days of course 1, patients undergo radiation therapy over 32-35 on weeks 1, 3, 5, 7 and 9.

After completion of study treatment, patients are followed up every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

- Localized urothelial cancer of bladder with presence of transitional cell carcinoma (TCC) component; mixed histologies are allowed Clinical or pathologic stage T2 -T4 disease including T4a and 4b if feasible to treat with radiation therapy Locoregional lymph node metastases are permitted but patients with distant metastases are ineligible; imaging to evaluate for distant metastases should consist of a minimum of computed tomography (CT)/magnetic resonance imaging (MRI) of abdomen/pelvis or CT urogram and a chest x-ray (CXR) or CT chest; patients for which there is clinical suspicion or symptoms of bone metastasis should have a bone scan completed to rule out metastatic disease prior to enrollment on study Agreeable to consider radiation therapy (RT) for the urothelial cancer: patients have to be evaluated by a radiation oncologist and deemed to be candidates for RT

The patients must not be candidates for chemotherapy due to at least one of the following reasons:

* Performance status of 2
* Creatinine clearance =< 60 ml/min as calculated by the Cockcroft-Gault formula
* Cardiac disease such as New York Heart Association (NYHA) class III or IV heart failure or cardiac ischemia within the last 12 months, grade 2 or greater neuropathy, or other comorbidities based on which patient is not considered a candidate for chemotherapy Alkaline phosphatase =< 3 x upper limit of normal Aspartate aminotransferase (AST) =< 3 x upper limit of normal Alanine aminotransferase (ALT) =< 3 x upper limit of normal Bilirubin < 1.5 x upper limit of normal (ULN) Absolute neutrophil count >= 1500/mm^3 Hemoglobin >= 9 g/dL Platelets >= 100 K/mm^3 Performance score (PS) of 0-2 by Zubrod score Life expectancy of 12 months Willingness to sign informed consent Patients cannot have active autoimmune disease or immunosuppressive conditions Serum creatinine =< 1.5 X institutional ULN or creatinine clearance > 40 ml/min as calculated by the Cockcroft-Gault formula In females with childbearing potential, or men with partners of child bearing potential, willingness to use adequate contraception for a minimum duration of 155 days in females and 215 days in males, after last dose of nivolumab Maximal tumor resection has been performed as feasible

Exclusion Criteria:

- The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) for urothelial cancer within 4 weeks, or intravesical Bacillus Calmette-Guerin (BCG) within 6 weeks of the first dose of study treatment Prior treatment with any PD-1 or PDL-1 inhibitor

The subject has received therapeutic radiation:

* To the bladder/prostate/rectum pelvis
* To any other site(s) within 28 days of the first dose of study treatment Obstructive renal failure that is not relieved with stents or nephrostomy tube/s The subject has received any other type of investigational agent within 28 days before the first dose of study treatment Steroid doses greater than an equivalent of prednisone 10 mg daily The subject has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test results at screening >= 2 x the laboratory ULN Uncontrolled hematuria

The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

* Cardiovascular disorders such as uncontrolled arrhythmias or uncontrolled congestive heart failure
* Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

  * Any of the following at the time of screening

    * Active peptic ulcer disease,
    * Active inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
  * Any of the following within 6 months before the first dose of study treatment:

    * History of abdominal fistula
    * Bowel perforation The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee Presence of another invasive malignancy, which required systemic therapy within 12 months of protocol enrollment, except for resected skin cancers or prostate cancer that is in remission Pregnant or nursing women Patient is a candidate for radical cystectomy as a potentially curative option. The patient may not be a candidate for radical cystectomy due to any of the following reasons: comorbidities, patient preference, or physician discretion. Patients with inherited syndromes associated with hypersensitivity to ionizing radiation (e.g., ataxia-telangiectasia, Nijmegen breakage syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 78.5 [54 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status Scale. Grade 0 to 5. 0=Normal activity, 1=Symptoms but ambulatory, 2=In bed <50% of the time, 3=In bed >50% of the time, 4=100% bedridden, 5=Dead
  Participants
    0 | 3
    1 | 16
    2 | 1
Pathological stage [Count of Participants; unit: Participants] — Pathologic stage T2 -T4 disease including T4a and 4b T2: tumor has spread to the muscle layer. T3: tumor invades the peripelvic fat, renal parenchyma, or into the fat around the ureter.
  T4: tumor invades nearby organs or outer layer of fat on the kidney. T4a: tumor invades the prostate, seminal vesicles, uterus, or vagina T4b: tumor has spread to the pelvic wall or the abdominal wall
  Participants
    T2Nx: Clinically main tumor invades muscularis propria, Cancer in lymph nodes cannot be measured. | 6
    pT2: Pathologically invades muscularis propria | 3
    pT2N1: Pathologically invades muscularis propria with a single node in the true pelvis | 1
    pT2Nx: Pathologically tumor invades muscularis propria, Cancer in lymph nodes not measurable. | 6
    pT2b: Pathologically invades the outer half of the muscularis propria. | 2
    pT4: Pathologically directly invades into adjacent structures. | 2
Prior Bacillus Calmette-Guerin (BCG) Therapy [Count of Participants; unit: Participants]
  No | 15
  Yes | 5
Prior Chemotherapy [Count of Participants; unit: Participants]
  No | 17
  Yes | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS distribution will be summarized with the Kaplan-Meier (K-M) survivorship estimate. A graph of the K-M curve for PFS will be generated along with the Hall-Wellner 90% confidence band, and a display of the number of patients at risk at several time points, below the X-axis. Summary statistics (12-month PFS rate, median PFS, etc.) will be calculated from the K-M life table, each one with its respective 90% confidence interval (CI).
Time Frame: From date of registration to date of first documented disease relapse/progression, or death from urothelial cancer whichever occurs first, assessed up to 12 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Number analyzed (Participants) | 20
months | 11.4 [7.5 to 23.7]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR will be estimated among all patients. Frequency distributions of best response will be generated. The point estimate of the ORR will be computed, along with its 95% (Wilson type) CI.
Time Frame: Up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage of response at 12 months
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Number analyzed (Participants) | 20
percentage of response at 12 months | 65.0 [43.3 to 81.8]

3. Secondary Outcome: Metastasis-free Survival (MFS)
Description: MFS will be calculated as a rate at 1 year with a 90% confidence interval from the K-M life tables.
Time Frame: From registration to the appearance of metastases or cancer related death, assessed up to 12 months
Measure: Number (90% Confidence Interval); unit: % of patients metastases-free at 1 year
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Number analyzed (Participants) | 20
% of patients metastases-free at 1 year | 63 [41 to 84]

4. Secondary Outcome: Overall Survival (OS)
Description: Summary statistics of OS will be calculated from the K-M life tables. K-M graphs of the censored OS distributions will also be generated.
Time Frame: From date of registration to death or last follow up, assessed up to 36 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Number analyzed (Participants) | 20
months | 15.6 [9.1 to 26.1]

5. Secondary Outcome: Quality of Life (QOL) and Bladder Functioning Questionnaires Assessment
Description: The QOL score will be measured pre therapy, during therapy and after therapy to compare the changes.
Time Frame: Up to 12 months
Population: Measure not taken
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: PD-1 and PDL-1 Expression Analysis Using Immunohistochemistry (IHC)
Description: PD-1 status will be checked on pre-therapy tumor tissue and will be correlated with the primary endpoint. Also, the PDL-1 status will be checked on pre-therapy tumor tissue and will be correlated with the primary endpoint.
Time Frame: Up to 12 months
Population: Those patients that had pre-therapy tumor tissue analyzed for PD-1 and PD-L1 (18 participants total).
Measure: Number (90% Confidence Interval); unit: % of patients progression-free at 1 year
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Number analyzed (Participants) | 18
% of patients progression-free at 1 year
  PD-1 <5: number analyzed (Participants) | 15
  PD-1 <5 | 44 [16 to 73]
  PD-1 =>5: number analyzed (Participants) | 3
  PD-1 =>5 | 35 [0 to 80]
  PD-L1 <5: number analyzed (Participants) | 12
  PD-L1 <5 | 36 [11 to 62]
  PD-L1 =>5: number analyzed (Participants) | 6
  PD-L1 =>5 | 55 [14 to 95]

7. Secondary Outcome: Th1/Th2 Cytokine Ratio Analysis
Description: The continuous markers (e.g., tumor infiltrating lymphocyte [TIL]s, Th1/Th2 cytokine ratio, etc.) will be summarized with standard descriptive statistics. These descriptive analyses of the serum markers will be performed for each time point at which the each marker is determined. Response (CR/PR vs not) will be modeled as a function of a dichotomized version of pre-study the continuous (ungrouped) markers (e.g., TILs from tissue, and the Th1/Th2 cytokine ratio from serum). The statistical goal of these exploratory analyses is to obtain the point and 95% CI estimates of the OR, and to simply determine the direction and approximate magnitude of these associations for use in planning a subsequent study. Censored PFS will be modeled as a function of a dichotomized version of the continuous (ungrouped) markers (e.g., TILs from tissue, and the Th1/Th2 cytokine ratio using Cox modelling strategy.
Time Frame: Up to 12 months
Population: Measure not taken
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed up to 36 months, and serious and Other (Not Including Serious) Adverse Events were assessed for up to 6 months
Arm/Group | Treatment (Nivolumab, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 13/20
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Radiation Therapy) (N=20)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Lymphocyte count decreased (Investigations) | 4 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (3)
Stroke (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Radiation Therapy) (N=20)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4)
Allergic reaction (Immune system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 6 (8)
Anxiety (Psychiatric disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (19)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Fatigue (General disorders) | 15 (18)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6)
Hypothyroidism (Endocrine disorders) | 2 (3)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (16)
Memory impairment (Nervous system disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Pain (General disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Platelet count decreased (Investigations) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 (5)
Sinusitis (Infections and infestations) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 5 (5)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (8)
Vaginal pain (Reproductive system and breast disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (4)
Weight loss (Investigations) | 1 (2)
Bladder spasm (Renal and urinary disorders) | 1 (2)
White blood cell decreased (Investigations) | 4 (4)
Edema limbs (General disorders) | 6 (7)
Infusion related reaction (General disorders) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT03421652/Prot_SAP_000.pdf